CLINICAL TRIAL: NCT02651753
Title: A Randomized, Open-label, Single Oral Dose, 2-way Crossover Clinical Trial to Compare Safety and Pharmacokinetic Characteristics of CKD-337 in Healthy Male Volunteers.
Brief Title: A Clinical Trial to Compare Safety and Pharmacokinetic Characteristics of CKD-337
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146BE15025
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin; Fenofibrate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Period 1: Reference drug (Lipitor+ Lipidil supra), 2 tablets administered under fed conditions.
  Period 2: Test drug(CKD-337), 1 capsule administered under fed conditions.
  Interventions: Drug: Lipitor + Lipidil supra; Drug: CKD-337
- B (Experimental): Period 1: Test drug(CKD-337), 1 capsule administered under fed conditions. Period 2: Reference drug (Lipitor+ Lipidil supra), 2 tablets administered under fed conditions.
  Interventions: Drug: Lipitor + Lipidil supra; Drug: CKD-337

INTERVENTIONS:
Drug: Lipitor + Lipidil supra — Reference Drug: Lipitor + Lipidil supra
  Other Names: Lipitor(Atorvastatin calcium trihydrate 21.70mg/tablet) + Lipidil supra(Fenofibrate 160mg/tablet)
Drug: CKD-337 — Test Drug: CKD-337
  Other Names: CKD-337(Atorvastatin calcium trihydrate 21.70mg+Cholinfe fenofibrate 178.8mg/capsule)

SUMMARY:
This study is a randomized, open-label, single oral dose, 2-way crossover clinical trial to compare safety and pharmacokinetics of CKD-337 in healthy male volunteers.

DETAILED DESCRIPTION:
This study is a randomized, open-label, single oral dose, 2-way crossover clinical trial to compare safety and pharmacokinetics of CKD-337 in healthy male volunteers.

Subjects will receive either a single oral dose of the test formulation(CKD-337) or a oral dose of the reference formulation(Lipitor+Lipidil supra).

Each treatment period was separated by a washout period of at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male older than 19 years at the time of screening
2. BMI 17.5~30.5 kg/m2 and body weight more than 55kg
3. Subject who is no chronic disease, no symptoms or pathological findings
4. Suitable subject who is determined by laboratory tests(hematology test, blood chemistry, urinalysis test) according to the characteristics of the drug and ECG test at the time of screening
5. Subject who fully understand the clinical trials after in-depth explanation, decided to join the clinical trials by their will and signed inform consent

Exclusion Criteria:

1. Subject who has a history of hepatic, kidneys, neurological, respiratory, endocrine, hemato-oncology, urinary, cardiovascular, musculoskeletal or psychiatric diseases that is clinically significant and who has a following history 1) Gallbladder disease including cholelithiasis, severe hepatic impairment 2) Acute/chronic pancreatitis due to hypertriglyceridemia 3) Pulmonary embolism or interstitial lung disease 4) Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption 5) Hypoalbuminemia 6) Alcoholics 7) Predisposition to rhabdomyolysis
2. Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption
3. Subject who has hypersensitivity to the drug composition containing choline fenofibrate, fenofibrate or atorvastatin, and other drug(aspirin, fenofibrate series, antibiotic and so on)
4. The following clinical significant findings at the time of screening

   * QTc > 450ms
   * PR interval > 200msec
   * QRS duration > 120msec
5. The following results in the clinical laboratory tests

   * CPK > 2 x upper limit of normal range
   * Liver function test (AST, ALT, ALP, Total bilirubin, γ-GT) > 2 x upper limit of normal range
   * eGFR(estimated GFR) < 60 mL/min/1.73m2
6. Systolic blood pressure ≥ 160mmHg or ≤ 100mmHg, Diastolic blood pressure ≥ 95mmHg or ≤ 60mmHg at the time of screening
7. History of drug abuse or a positive reaction for drug abuse at the screening test for urine
8. Taking ETC, oriental medicine within 2 weeks and OTC, vitamin within 1 week before the first dosing
9. Taking the medication involved in other clinical trials within 3 months before the first dosing
10. Whole blood donation with 2 months or component blood donation within 1 month or blood transfusion within 1 month before the first dosing
11. Alcohol > 21 units/week (1unit=10g of pure alcohol), within 6 month before the first dosing
12. Smoker(> 10 cigarettes/day) for the last 3 months
13. Comsumption of grapefruit of food containing grapefruit during clinical trial period from first dosing 48hours ago
14. Comsumption of food containing caffeine(e.g. coffee, green tea) during 24 hours ago IP dosing at discharge
15. Not using a reliable contraception, planning a pregnancy during the study
16. An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Atorvastatin AUCt | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin Cmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Fenofibric acid AUCt | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Cmax | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration

SECONDARY OUTCOMES:
Atorvastatin AUCinf | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin Tmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin t1/2 | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin CL/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin Vd/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Fenofibric acid AUCinf | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Tmax | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid t1/2 | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid CL/F | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Vd/F | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
2-hydroxy atorvastatin AUCt | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Cmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin AUCinf | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Tmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin t1/2 | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin CL/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Vd/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration

IPD SHARING:
Plan to Share IPD: No